CLINICAL TRIAL: NCT00912691
Title: A Phase III Open Label Extension Study of CM-AT in Children With Autism
Brief Title: A Trial of CM-AT in Children With Autism- Open Label Extension Study
Acronym: CM-AT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Curemark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00102/Autism
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Autism
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): CM-AT
  Interventions: Drug: CM-AT

INTERVENTIONS:
Drug: CM-AT — Single unit dose powder of active substance (CM-AT) administered 3 times per day for 90 days

SUMMARY:
The purpose of this study is to determine whether CM-AT is effective in treating the core symptoms of autism.

DETAILED DESCRIPTION:
Autism is currently a significant cause of disability in the pediatric population. CM-AT is based upon the observation that many children with autism do not digest protein. CM-AT is a proprietary enzyme that is designed as a powder taken three times a day. It is formulated to be released in the small intestine to enhance protein digestion thus increasing the availability of essential amino acids.

ELIGIBILITY:
Inclusion Criteria:

* Meets the current Diagnostic and Statistical Manual for Mental Disorders (DSM-IV-TR) diagnostic criteria for autistic disorder (AD)
* Ongoing 00102 Protocol required completion of 00101 Protocol
* Now recruiting subjects directly into 00102 Protocol

Exclusion Criteria:

* Ongoing study required patients to be 3-8 years old weighing < 11kg (24.2 lbs.), and achieving ages 9-12 years old weighing < 22kg (48.4 lbs.).
* Newly recruited subjects must be between ages 9 - 12 years old weighing < 22kgs (48.4 lbs.)
* Demonstrated previous allergy to porcine (pork) products
* Previous history of severe head trauma or stroke, seizure within one year of entering study or uncontrolled systemic disease
* Diagnosis of: HIV, cerebral palsy, endocrine disorder, pancreatic disease
* Within 30 days of starting the study, certain supplementation, chelation or dietary restriction (a 30 day washout period would be required for inclusion)
* Any use of psychotropic medications, stimulants, or SSRI's must be discontinued for 30 days prior to entrance

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Evidence of changes in behavior scales associated with the core symptoms of autism | Baseline, 4, 8, 12, 16, 20, 24, 36, 60, 72, 84,96,108,120,132,144,156, 168, and 180 weeks

SECONDARY OUTCOMES:
Other key measures of behavior and quality of life associated with autism | Baseline, 4, 8,12,16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Arnold, MD, Principal Investigator — Ohio State University, Nisonger Center
Locations (19):
- United States (19):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - University of California, Davis, M.I.N.D. Institute, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Lake Mary Pediatrics, Orange City, Florida
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Louisiana State University, Shreveport, Louisiana
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Mount Sinai School of Medicine, Manhattan, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oklahoma State University, Child Study Center, Oklahoma City, Oklahoma
  - Cyn3rgy Research Center, Gresham, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Universtiy of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Houston, Houston, Texas
  - Ericksen Research & Development, Clinton, Utah